CLINICAL TRIAL: NCT07388589
Title: The Soluble and Osmotic Fibre (SOLOS) Diet for Functional Bowel Disorders With Constipation
Brief Title: Soluble and Osmotic Fibre (SOLOS) Diet for Constipation
Acronym: SOLOS
Status: Not yet recruiting | Type: Observational
Sponsor: Singapore Institute of Technology (Other)
Responsible Party: Principal Investigator, Wilson Bridgette Jane, Assistant Professor, Singapore Institute of Technology
Other Study IDs: RECAS-0723-IRB
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Constipation; Constipation - Functional; Constipation Chronic Idiopathic; Constipation Predominant Irritable Bowel Syndrome; Constipation, Signs and Symptoms, Digestive; Constipation-predominant IBS (IBS-C); Constipation-predominant Irritable Bowel Syndrome; Constipation-predominant Irritable Bowel Syndrome (IBS-C); Diet Therapy; Diet Modification; Diet, Food and Nutrition; Dietary and Nutritional Therapies; Dietary Fiber; Dietary Fibers
Keywords: Constipation; Functional constipation; Constipation-predominant irritable bowel syndrome (IBS-C); Soluble fiber; osmotic sugar
MeSH Terms: conditions — Constipation | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Functional Constipation
  Interventions: Other: Diet
- Patients with IBS-C or SIBO-C
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Dietary advice combining increased intake of dietary sources of soluble fibres and osmotic sugars in improving constipation symptoms.
  Other Names: soluble fibre and osmotic carbohydrates diet; soluble fibre and osmotic carbohydrates (SOLOS) diet; SOLOS diet

SUMMARY:
This research aims to study the dual effectiveness of incorporating soluble fibre and osmotic carbohydrates (SOLOS), with or without restricting fructans and GOS, and present novel findings in managing GI symptoms in patients with functional bowel disorders with constipation. These findings may also support researchers and clinicians in shaping new dietary approaches in the management of general constipation symptoms.

DETAILED DESCRIPTION:
Aims: This retrospective clinical audit study aims to evaluate the effectiveness of dietary advice promoting increased intake of soluble fibre and poorly absorbed (osmotic) carbohydrates, with or without restriction of fructans and galacto-oligosaccharides (GOS), on adult patients (18-70 years old) with functional bowel disorders with constipation from the UK by comparing to baseline scores for severity and frequency of gastrointestinal symptoms and stool output.

Hypothesis: The dietary advice promoting increased intake of soluble fibre and osmotic sugars will produce a significant change from baseline in gastrointestinal symptoms and stool output in adult patients (18-70 years old) with functional bowel disorders with constipation from the UK.

Methodology: The study population will include all patients who have consulted with the Principal Investigator, a specialist gastroenterology dietitian between January 2021 and December 2025. All patients who have met the inclusion criteria will then form the research sample. Eligible subjects' data and study variables will be extracted from patient letters and clinical management records without direct patient contact. These study variables include the frequency and severity of the patients' symptoms at their initial appointment and follow-up appointment if available. Anthropometric data such as height and weight will also be obtained. The compiled data will then be analysed by conducting statistical tests, specifically the paired t-test, which will produce descriptive statistics that will interpret the effectiveness of the SOLOS diet on patients with functional bowel disorders with constipation.

Applications: To date, there has not been any study studying the dual effects of soluble fibre and osmotic carbohydrates consumption on alleviating constipation-related symptoms in patients with functional bowel disorders with constipation. Therefore, this research aims to present novel findings that can advance existing dietary management of functional bowel disorders with constipation. These results are expected to deepen understanding and research in food manufacturing and clinical nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Presented with symptoms of FC, IBS-C, or SIBO-C
* Were aged 18 to 70 years old. (Research focus is on adult patients, excluding older adults and children)
* Date of baseline (first) and follow-up appointments ranged from January 2021 to December 2025
* Did not attend follow-up appointments (Data would be treated as "intention to treat" and data points were carried forward for conservative analysis).

Exclusion Criteria:

* Had no history of constipation-related symptoms (Does not relate to research question's population or outcome)
* Started treatment before January 2021
* Were not due for follow-up before the end of December 2025
* Symptom and stool data inadequately recorded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-70 years old) with functional bowel disorders with constipation from the UK, seen by a specialist dietitian (Principal Investigator)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Stool frequency | January 2021 to December 2025
  Frequency of stool output per week
Stool form | January 2021 to December 2025
  Bristol Stool Form Scale
Gastrointestinal Symptom Frequency | January 2021 to December 2025
  Frequency of gastrointestinal symptom in a week, recorded as number of days out of 7 the symptom occurred over the past week.
Gastrointestinal Symptom Severity | January 2021 to December 2025
  Severity of symptoms in a week scored using Gastrointestinal Symptom Rating Scale (GSRS). Scores range from 0 (absent) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette J Wilson, Dr, Principal Investigator — Singapore Institute of Technology
Locations (1):
- Singapore Institute of Technology, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided